CLINICAL TRIAL: NCT05463796
Title: InAdvance: Surveillance, Prevention, and Interception in a Population at Risk For Cancer
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Sapna Syngal, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 22-200
Record Dates: First submitted 2022-06-24; First posted 2022-07-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer Risk; Cancer Predisposition Syndrome; Hereditary Cancer Prediction; Childhood Cancer Survivors; Adult Cancer Survivors; IARC Carcinogens; Smoking History; Lung Cancer; Ductal/Lobular Carcinoma; Barrett Esophagus; Pancreatic Precursor Lesions; Colonic Dysplasia/Adenomata; Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis; Cirrhosis; High Grade Prostatic Epithelial Neoplasia; High-grade Bladder Urothelial Dysplasia/Carcinoma in Situ; Adenomatous Hyperplasia; High-risk Oral Precancerous Diseases; Melanocytic Lesion, Adult; Hematologic Malignancy; Lung; Node; Serous Tubal Intraepithelial Carcinoma; Endometrial Intraepithelial Neoplasia; Cervical and Endocervical Carcinoma in Situ; Vulvar Intraepithelial Neoplasia; Nephrogenic Rests; Benign Bone Lesions With Risk of Malignant Degeneration; Giant Cell Tumor; Osteochondroma; Spitz Nevus
Keywords: Hereditary Risk for Cancer; Childhood cancer survivors; Adult cancer survivors; Precursor Lesions
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Lobular; Barrett Esophagus; Non-alcoholic Fatty Liver Disease; Fibrosis; Carcinoma in Situ; Hematologic Neoplasms; Endometrial Hyperplasia; Giant Cell Tumors; Osteochondroma; Nevus, Epithelioid and Spindle Cell | interventions — Sampling Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Patients' specimens including blood, buccal swab or mouthwash, urine, stool, bone marrow, tissue from biopsy or surgical excision, bodily fluids or other specimens will be collected from patients who consent to the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- HEREDITARY RISK: Participants will also be asked to complete an intake survey that will include questions about demographics, medical history and family history data.
  Tissue samples will be collected during a routine visit.
  Participants will be asked to donate any of the following tissue types:
  * Blood
  * Buccal swab (saliva) or mouthwash
  * Urine
  * Stool
  * Biopsy or surgical tissue (i.e., bone marrow)
  * Bodily fluids
  * Other tissues
  Interventions: Other: Samples
- EXPOSED HIGH RISK: Participants will also be asked to complete an intake survey that will include questions about demographics, medical history and family history data.
  Tissue samples will be collected during a routine visit.
  Participants will be asked to donate any of the following tissue types:
  * Blood
  * Buccal swab (saliva) or mouthwash
  * Urine
  * Stool
  * Biopsy or surgical tissue (i.e., bone marrow)
  * Bodily fluids
  * Other tissues
  Interventions: Other: Samples
- PRECURSOR LESIONS: Participants will also be asked to complete an intake survey that will include questions about demographics, medical history and family history data.
  Tissue samples will be collected during a routine visit.
  Participants will be asked to donate any of the following tissue types:
  * Blood
  * Buccal swab (saliva) or mouthwash
  * Urine
  * Stool
  * Biopsy or surgical tissue (i.e., bone marrow)
  * Bodily fluids
  * Other tissues
  Interventions: Other: Samples
- FAMILY MEMBERS: These family members will be identified by the patients participating in the study. Blood, buccal cells, or saliva or oral rinses will be collected in one of three ways from family members of patients (i) at the time of consent; (ii) via a mailed blood kit or saliva kit; or (iii) at a separate appointment scheduled by the consented participant
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Tissue samples will be collected during a routine visit. Participants will be asked to donate any of the following tissue types:
  Blood, Buccal swab (saliva) or mouthwash, Urine, Stool, Biopsy or surgical tissue (i.e., bone marrow),Bodily fluids, Other tissues

SUMMARY:
This research study is creating a way to collect and store specimens and information from participants who may be at an increased risk of developing cancer, or has been diagnosed with an early phase of a cancer or a family member who has a family member with a precursor condition for cancer.

* The objective of this study is to identify exposures as well as clinical, molecular, and pathological changes that can be used to predict early development of cancer, malignant transformation, and risks of progression to symptomatic cancer that can ultimately be fatal.
* The ultimate goal is to identify novel markers of early detection and risk stratification to drive potential therapeutic approaches to intercept progression to cancer.

DETAILED DESCRIPTION:
The objective of this protocol is to obtain clinical information and facilitate the collection and distribution of specimens obtained during the course of clinical care or research participation.

* Blood, buccal swabs, urine or tissue or other body fluids (including stool) may be specifically acquired for research in order to perform molecular and other types of analyses for research purposes.
* These materials will be collected from all eligible participants who have a precursor lesion or an increased risk of cancer

It is expected that about 5,000 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants to be included in this study include the following (note that this list is not comprehensive but gives examples of precursor conditions for each organ type):

  1-Hereditary risk for cancer including
  * Carriers of known or previously unrecognized pathogenic germline variants of cancer predisposing genes
  * Individuals with personal or family history suggestive of elevated cancer risk (this may include individuals who have negative genetic testing results or have not elected to undergo testing)
  * Individuals with a clinically based diagnosis of a Cancer Predisposition Syndrome (examples, neurofibromatosis, Fanconi Anemia, Ataxia-Telangiectasia)
  * Hereditary Cancer Prediction Model-based elevated cancer risk
  * Others at risk for specific cancers by virtue of exposure, obesity, gender, race and ethnicity, HPV exposure (for H&N cancer for example), etc.
* Exposed High Risk including

  * Childhood cancer survivors with treatment exposures associated with increased risk of cancer
  * Adult cancer survivors with treatment exposures associated with increased risk of cancer
  * Documented high level exposure to group 1 IARC carcinogens
  * Thoracic: individuals at risk for lung cancer including but not exclusive of the following criteria: Age >50, Smoking history of >15 pack years, First-degree relative history of lung cancer or COPD
  * alcoholic liver disease (NAFL), non-alcoholic steatohepatitis (NASH), cirrhosis
* Precursor Lesions including

  * Breast: ductal/lobular carcinoma in situ (CIS) and atypical hyperplasia
  * GI: Barrett's esophagus, Pancreatic precursor lesions, colonic dysplasia/adenomata, nonalcoholic fatty liver (NAFL), nonalcoholic steatohepatitis (NASH), cirrhosis
  * GU: High grade prostatic epithelial neoplasia, and high-grade bladder urothelial dysplasia/carcinoma in situ,
  * Lung: Adenomatous hyperplasia
  * H&N: high-risk oral precancerous diseases
  * Skin: Class II melanocytic lesions. Squamous dysplasia
  * Heme malignancies: CHIP, CCUS, ICUS, MGUS, SMM, SWM, MBL (spell these out), Low grade lymphomas
  * Thoracic: Lung nodules detected on screening CT that prompt further follow-up
  * GYN: STIC lesion (serous tubal intraepithelial carcinoma), Endometrial intraepithelial neoplasia, Cervical and endocervical carcinoma in situ, vulvar intraepithelial neoplasia
  * Pediatric histologic diagnoses sometimes associated with development of malignancy: Nephrogenic rests, benign bone lesions with risk of malignant degeneration (Giant cell tumor, osteochondroma), Spitz nevus, and others.
* FAMILY MEMBERS or healthy individuals

Exclusion Criteria:

There are no exclusion criteria for the study.

Note: Patients with prior cancer history are allowed to participate. Patients with prior history of cancer or non-metastatic localized cancers (such as skin cancer or localized prostate cancer) are allowed to be enrolled. Patients enrolled in clinical trials or receiving therapy for precursor diseases are NOT excluded from this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants to be included in this study include the following (note that this list is not comprehensive but gives examples of precursor conditions for each organ type Hereditary risk for cancer, Exposed High Risk, Precursor Lesions, FAMILY MEMBERS
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2032-03-25 (Estimated)

PRIMARY OUTCOMES:
Identify exposures as well as clinical, molecular, and pathological changes that can be used to predict early development of cancer, malignant transformation, and risks of progression to symptomatic cancer that can ultimately be fatal. | 5 years
  The InAdvance Study will screen participants for precancerous conditions and cancer through blood tests and tissue biopsies. These biologic samples will be screened for precancerous conditions through routine clinical methods, as well as using novel research level technology. This could include germline testing, whole genome and whole exome sequencing. The participants will be followed serially to track their disease progression. Participants will fill out general health questionnaires, and we will match their answers to the timepoint of their sample submission and follow changes to their answers.

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Syngal, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu